CLINICAL TRIAL: NCT01767740
Title: Two-Arm, Single Blind, Randomized Pilot Study on the Use of ULTRABRAID PLUS SUTURE in the Repair of Tears of the Rotator Cuff
Brief Title: Pilot Study of the Use of ULTRABRAID PLUS SUTURE in the Repair of Tears of the Rotator Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15001105
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Supraspinatus Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ULTRABRAID PLUS SUTURE (Experimental): ULTRABRAID Plus Suture manufactured by Smith & Nephew used in subjects undergoing rotator cuff repair.
  Interventions: Device: ULTRABRAID PLUS SUTURE
- ULTRABRAID SUTURE (Active Comparator): ULTRABRAID Suture is a marketed suture manufactured by Smith & Nephew used in subjects undergoing rotator cuff repair.
  Interventions: Device: ULTRABRAID SUTURE

INTERVENTIONS:
Device: ULTRABRAID PLUS SUTURE — Rotator Cuff Repair with ULTRABRAID PLUS SUTURE
  Arms: ULTRABRAID PLUS SUTURE
Device: ULTRABRAID SUTURE — Rotator Cuff Repair with ULTRABRAID SUTURE
  Arms: ULTRABRAID SUTURE

SUMMARY:
The primary objective of this study is to obtain safety data on the use of the ULTRABRAID PLUS SUTURE, and to assess the preliminary effectiveness of the use of the ULTRABRAID PLUS SUTURE in comparison to the ULTRABRAID SUTURE in patients undergoing rotator cuff repair.

DETAILED DESCRIPTION:
The primary objective of this two-arm, randomized, single-blind pilot study is to obtain safety data on the use of the ULTRABRAID Plus Suture and to assess the preliminary effectiveness of the use of the ULTRABRAID Plus Suture in comparison to the ULTRABRAID Suture in subjects undergoing rotator cuff repair. The primary endpoint of the 6-month postoperative analysis is to assess rotator cuff integrity at 6 months, defined as the proportion of subjects with a re-tear of the rotator cuff as measured by high-resolution ultrasound.

Secondary endpoints include:

rotator cuff integrity at the other time points, as well as between arms (1, 3, 6 weeks and 3, 12 months); difference in tissue thickness and muscle atrophy using high-resolution ultrasound between baseline (preoperative) and all postoperative time points (1, 3, 6 weeks and 3, 6, 12 months); difference in tendon echogenicity and vascularity using Doppler ultrasound between baseline (preoperative) and all postoperative time points (1, 3, 6 weeks and 3, 6, 12 months); difference in Constant Shoulder Assessment score and Western Ontario Rotator Cuff (WORC) Index between baseline (preoperative) and all postoperative time points (1, 3, 6 weeks and 3, 6, 12 months); rehabilitation:

* time to active-assisted rehab exercises
* time to isometric rehab exercises
* time to discontinuation of an arm sling lab results (C-Reactive Protein [CRP], Erythrocyte Sedimentation Rate [ESR] and Butyric Acid Levels) at 1, 3, and 6 weeks postoperatively; adverse event (AE) rates (all categories).

ELIGIBILITY:
Inclusion Criteria (Subjects must meet ALL of the following criteria):

* Male or female, aged 18 to 70 years at the time of surgery
* Willing and able to give voluntary informed consent to participate in this investigation
* Small (<1cm), Medium (1-3cm) or large (>3-5cm) tear of the supraspinatus tendon, which may or may not include the infraspinatus tendon of the rotator cuff. Tear size will be based on area of longest dimension as evidenced by clinical examination and diagnostic imaging prior to surgery, with the definitive measurement confirmed at surgery
* Tear requires repair within two years of initial diagnosis
* Tear must be anatomically repairable (must be able to get tendon back to the medial position on the footprint and at least back to the tuberosity)
* Willing and able, in the opinion of the Investigator, to cooperate with study procedures, and willing to return to study site for physical therapy and all post-operative study visits

Exclusion Criteria (Subjects must not meet ANY of the following criteria):

* Tears involving tendons other than the supraspinatus and infraspinatus
* Partial thickness tears of the rotator cuff (tear must be full thickness)
* Evidence of acute trauma including fracture or dislocation of the shoulder joint
* Chronic retraction
* Evidence of active infection, osteomyelitis, sepsis or distant infection which could spread to the index joint
* Subject has had previous rotator cuff, arthroplasty or fracture procedures on the operative shoulder
* Subject has had acromioplasty or diagnostic arthroscopy on the operative shoulder within one (1) year prior to scheduled surgery date
* Evidence of osteomalacia or other metabolic bone disorder(s) which may impair bone or soft tissue function
* Evidence of other significant shoulder pathology including (Type II-IV lesion, Bankart lesion, Hill Sachs lesion)
* Patient has grade 4 changes to articular cartilage in operative shoulder
* Inflammatory arthropathies
* Significant muscle paralysis of the shoulder girdle.
* Painful pathologies of the cervical spine
* Comminuted bone surface, which would compromise secure anchor fixation.
* Subject has a known sensitivity to implant materials, including sodium butyrate.
* Non-surgical rotator cuff associated treatment, such as corticosteroid injection, within one (1) month prior to scheduled surgery date
* Participating in another investigational trial or ongoing study that would interfere with the assessment of the primary and secondary outcomes
* Female patient who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods
* Currently known to abuse drugs or alcohol which could affect follow-up care or treatment outcomes
* Current smoker
* Major psychiatric illness, developmental handicap or inability to read and understand the English language
* Major medical illness that would preclude undergoing surgery
* Known to be involved in any active injury litigation claims relating to the study shoulder
* Unwilling or unable to be assessed according to study protocol for one year following surgery
* Patient requires a concomitant SLAP repair procedure in operative shoulder
* Surgeon plans to use transosseous sutures in the study procedure
* Surgeon plans to use a Platelet Rich Plasma product or another therapy intended to augment healing of the rotator cuff in the study procedure
* Protocol specified surgical technique cannot be followed for this subject
* Rotator cuff repair will be done via open (as opposed to arthroscopic) procedure
* Any other reason (in the judgment of the investigator)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rotator Cuff Integrity | 6 months post-operatively
  The primary endpoint of the 6-month postoperative analysis is to assess rotator cuff integrity at 6 months, defined as the proportion of subjects with a re-tear of the rotator cuff as measured by high-resolution ultrasound.

SECONDARY OUTCOMES:
Rotator Cuff Integrity | 1, 3 and 6 weeks and 3 and 12 months post-operatively
  To assess rotator cuff integrity defined as the proportion of subjects with a re-tear of the rotator cuff as measured by high-resolution ultrasound.
Change in post-surgery tissue thickness, rotator cuff integrity, tendon echogenicity and muscle atrophy | 1, 3 and 6 weeks and 3, 6 and 12 months post-operatively
  Compared to Baseline (preop)
Change in Vascularity | 1, 3 and 6 weeks and 3, 6 and 12 months post-operatively
  Compared to Baseline (preop)
Change in Constant Shoulder Assessment | 1, 3 and 6 weeks and 3, 6 and 12 months post-operatively
  Compared to Baseline (preop)
Change in Western Ontario Rotator Cuff Index | 1, 3 and 6 weeks and 3, 6 and 12 months post-operatively
  Compared to Baseline (preop)
Rehabilitation | 3 and 6 weeks and 3, 6 and 12 months post-operatively
  * Time to active-assisted rehab exercises
  * Time to isometric rehab exercises
  * Time to discontinuation of arm sling
Labs | 1, 3 and 6 weeks (optional 3, 6 and 12 months) post-operatively
  Compared to Baseline (preop) Note: If levels do not return to baseline, tests will continue beyond 6 weeks
Adverse Events | Surgery and 1, 3 and 6 weeks and 3, 6 and 12 months post-operatively
  All AE measured and observed, from the initiation of the surgical procedure and throughout the subjects participation in the study, were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litchfield, MD, FRCSC, Principal Investigator — Fowler Kennedy Sports Medicine Clinic
Locations (4):
- Canada (4):
  - Innovation Science and Medicine, Burlington, Ontario
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - St. Josephs Hospital, London, Ontario
  - Women's College Hospital, Toronto, Ontario